CLINICAL TRIAL: NCT02580279
Title: Phase II Study of Topical Epigallocatechin-3-gallate (EGCG) in Patients With Breast Cancer Receiving Adjuvant Radiotherapy
Brief Title: Study of Epigallocatechin-3-gallate (EGCG) for Skin Prevention in Patients With Breast Cancer Receiving Adjuvant Radiotherapy
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Shandong Cancer Hospital and Institute (Other)
Responsible Party: Principal Investigator, Han Xi Zhao, Principal Investigator, Shandong Cancer Hospital and Institute
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: GTEBC-2015
Record Dates: First submitted 2015-09-27; First posted 2015-10-20 (Estimated); Last update posted 2019-04-05 (Actual); Status verified 2019-04

CONDITIONS: Breast Neoplasms; Dermatitis; Prevention & Control; Epigallocatechin Gallate
Keywords: Breast Neoplasms; prevention & control; Epigallocatechin gallate; Dermatitis
MeSH Terms: conditions — Breast Neoplasms; Dermatitis

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- EGCG group (Experimental): EGCG (purity≥95% by high pressure liquid chromatography; from Ningbo HEP Biotech Co., Ltd) is dissolved in 0.9% saline solution;The solution is sprayed three times a day at 0.05 ml/cm2 to the whole radiation field until two weeks after radiation completion; Patients who developed grade Ⅱ radiation-induced dermatitis have the option to either withdraw from the study or to continue with EGCG. Patients are follow general good skin care practices during radiation therapy, such as not applying water soaks to relieve itching or pain, not vigorously rubbing the irradiated area, or not erasing ink marks; patting the skin dry with a soft towel; avoiding exposure to the sun; and wearing loose and cotton clothes. They are advised not to use deodorant, lotion, cream, make up, perfume or any other product on the area during the course of radiation therapy.
  Interventions: Drug: EGCG
- placebo (Placebo Comparator): The placebo is 0.9% saline solution.Patients are also to follow general good skin care practices which is same as the EGCG group.
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: EGCG
  Arms: EGCG group
Drug: placebo
  Arms: placebo

SUMMARY:
The investigators conduct this phase II study of EGCG therapy protection of the skin from damage induced by radiotherapy in breast cancer. In order to observe the effectiveness of EGCG, investigators will utilize both clinician assessments and patient self-assessments. Physician's skin assessments will be scored utilizing the Radiation Therapy Oncology Group (RTOG) score. Patient reported symptom scores are adapted from the Skin Toxicity Assessment Tool (STAT) as pain, burning, itching, pulling, and tenderness in the treatment area. The scales are translated into Chinese and guides in Chinese are developed instructing how to use the scales and perform the assessments.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ eighteen years
* Eastern Cooperative Oncology Group performance status of 0-1
* Normal hematologic, hepatic function and renal values
* Forced expiratory volume 1 >800 cc

Exclusion Criteria:

* The presence of rash or unhealed wound in the radiation field
* A known allergy or hypersensitivity to EGCG
* Pregnancy or lactation
* History of/current connective tissue disorder
* Prior radiation to the thorax

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Estimated)
Dates: Start 2014-12; Primary Completion 2019-08 (Estimated); Study Completion 2019-10 (Estimated)

PRIMARY OUTCOMES:
Superiority of EGCG in reducing Grade II or more dermatitis as assessed by Radiation Therapy Oncology Group (RTOG) scores in patients with breast cancer receiving radiation | Each patient will be enrolled for a 5-6 week trial

SECONDARY OUTCOMES:
Superiority of EGCG in reducing pain as assessed by the Skin Toxicity Assessment Tool (STAT) in patients with breast cancer receiving radiation | Each patient will be enrolled for a 5-6 week trial
Improved quality of life with usage of EGCG for treatment of radiation-dermatitis in patient with breast cancer | Each patient will be enrolled for a 5-6 week trial
  questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Ligang Xing, MD,PhD, Study Chair — Shandong Cancer Hospital and Institute

REFERENCES:
- [Derived] Xie J, Jia L, Xie P, Yin X, Zhu W, Zhao H, Wang X, Meng X, Xing L, Zhao H, Li X. Efficacy and safety of epigallocatechin-3-gallate in treatment acute severe dermatitis in patients with cancer receiving radiotherapy: a phase I clinical trial. Sci Rep. 2023 Aug 24;13(1):13865. doi: 10.1038/s41598-023-40881-4. PMID 37620508
- [Derived] Zhao H, Zhu W, Zhao X, Li X, Zhou Z, Zheng M, Meng X, Kong L, Zhang S, He D, Xing L, Yu J. Efficacy of Epigallocatechin-3-Gallate in Preventing Dermatitis in Patients With Breast Cancer Receiving Postoperative Radiotherapy: A Double-Blind, Placebo-Controlled, Phase 2 Randomized Clinical Trial. JAMA Dermatol. 2022 Jul 1;158(7):779-786. doi: 10.1001/jamadermatol.2022.1736. PMID 35648426